CLINICAL TRIAL: NCT02501707
Title: The Value of Echocardiography for Prediction of Radiation-induced Lung Injury in Non-small Cell Lung Cancer Patients Treated With Chemoradiation: an Onco-cardiac Prospective Cohort Study.
Brief Title: Echocardiography for RILI Prediction
Status: Terminated | Type: Observational
Why Stopped: The study is prematurely terminated due to bad inclusion and the fact that examinations are already being used in standard care.
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Sponsor
Other Study IDs: echocardiographyRILI
Record Dates: First submitted 2015-07-13; First posted 2015-07-17 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: NSCLC
Keywords: echocardiography; radiation-induced lung injury; prognostic; chemo radiotherapy; non-small cell lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bloodsamples and saliva samples will be collected according to the biobank protocol at Maastro clinic to explore the prognostic value of mitochondrial DNA for development of radiation-induced lung injury.
  Cardiac bloodmarkers: B-type Natriuretic Peptide (BNP), cardiac Troponin I and T will be measured.
  Haemoglobin and inflammatory parameters (CRP, IL-6 and TNFa)
Oversight: Data Monitoring Committee: No

SUMMARY:
Severe radiation-induced lung injury (RILI) occurs in approximately 20% of the lung cancer patients, who are treated with curative chemoradiation. In this study the investigators want to evaluate the prognostic value of baseline cardiac function assessed with echocardiography for prediction of RILI.

DETAILED DESCRIPTION:
Severe radiation-induced lung injury (RILI) occurs in approximately 20% of the lung cancer patients, who are treated with curative chemoradiation (CRT).This side-effect can heavily impact quality of life and is a dose-limiting factor for the treatment. Identifying high risk patients before the start of the treatment would make it possible to adapt the treatment by choosing another radiation technique or proton therapy. However, despite the fact that many patient and treatment characteristics have been associated with RILI, it is not possible to accurately predict the risk of RILI for individual patients. Recently, it has been shown that the radiation dose to the heart is a risk factor for lung toxicity in both animal and clinical studies. Also, in a study, carried out jointly by CARIM and GROW, it was found that patients with a previous diagnosis of cardiac disease had a significantly higher risk to develop RILI after CRT (p-value <0.001), even with low or no radiation dose to the heart. It is unknown whether asymptomatic cardiac comorbidity is also related to development of RILI. Taking into account that approximately 30% of all lung cancer patients suffer from symptomatic cardiac comorbidity at the start of cancer treatment, there is an urgent need for research projects focusing on cardio-oncology. These projects will make it possible to unravel the complex relationship between heart, lungs, chemotherapy and radiation treatment. In the current project the investigators hypothesize that biomarkers based on echocardiography, which reflects cardiac function, are prognostic for development of radiation induced lung injury after chemoradiotherapy. In addition, the investigators will validate our previous finding that presence of cardiac comorbidity is associated with RILI.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage I-III non small cell lung cancer, excluding malignant pleural/pericardial effusion
* Planned for curatively intended primary (chemo)radiotherapy, due to irresectable disease and/or medical inoperability
* WHO performance status 0-2
* No history of prior chest radiotherapy
* No uncontrolled infectious disease
* No other active malignancy
* No prior lung surgery (VATS, wedge resection, segment resection, lobectomy)
* Willing and able to comply with the study prescriptions
* 18 years or older
* Ability to give and having given written informed consent before patient registration

Exclusion Criteria:

* malignant pleural/pericardial effusion
* history of prior chest radiotherapy
* uncontrolled infectious disease
* other active malignancy
* prior lung surgery (VATS, wedge resection, segment resection, lobectomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to MAASTRO Clinic with non-small cell lung cancer stage I-III disease can be included in this study (approximately 160 patients per year).
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Dyspnea score at three months after (chemo)radiotherapy, assessed by the patient version of the CTCv4.0 | up to 3 months

SECONDARY OUTCOMES:
Dyspnea score at six months after (chemo)radiotherapy, assessed by the patient version of CTCv4.0 | up to 6 months
Changes in dyspnea score after radiotherapy, compared to baseline | up to 12 months
Change in Left Ventricle Ejection Fraction (LVEF) (baseline versus 3-month after chemo radiation) | up to 3 months
Change in left atrial volume (2009 AHA/ESC guidelines)(baseline versus 3-month after chemo radiation) | up to 3 months
Radiation pneumonitis at 3-months after start of radio(chemo)therapy, assessed on a follow-up 3D CT scan image. | up to 3 months
Lung fibrosis score at 6-months after start of chemo radiation, assessed on a follow-up CT scan image | up to 6 months
Prevalence-based dyspnea measure, reflecting severity as well as duration of dyspnea | up to 12 months
Changes in physical activity levels and sedentary behavior, assessed by accelerometry | up to 12 months
Pulmonary function based on spirometry | up to 3 months
Change in left atrial ejection fraction (from pts in SR)(2009 AHA/ESC guidelines)(baseline versus 3-month after chemo radiation) | up to 3 months
Change in mitral inflow (2009 AHA/ESC guidelines)(baseline versus 3-month after chemo radiation) | up to 3 months
Change in pulmonary vein inflow patterns (2009 AHA/ESC guidelines)(baseline versus 3-month after chemo radiation) | up to 3 months
Change in tissue doppler patterns of the mitral annulus (2009 AHA/ESC guidelines)(baseline versus 3-month after chemo radiation) | up to 3 months
Cardiac blood biomarkers at baseline and during treatment, Brain natriuretic peptide(BNP), troponin I (TnI) and troponin T(TnT) | up to 3 months
Haemoglobin parameters in the blood at baseline and during treatment | up to 3 months
Inflammatory parameters (CRP, IL-6 and TNFa) in the blood at baseline and during treatment | up to 3 months
Time trends in physical activity and sedentary time from baseline till 12 months after radiotherapy, measured by accelerometers in four weekly periods | up to 12 months

OTHER OUTCOMES:
Cardiac Comorbidity according to ICD v10 | up to 12 months
Radiomics (the evolving field of texture analysis) of normal tissue(heart and lung) | up to 3 months
Mitochondrial DNA (prognostic value of mtDNA for development of RILI) | up to 12 months
Body composition, analysed by evaluation of muscle mass and fat mass on computed tomography (CT) scans at a standardized vertebral landmark (third lumbar vertebra) | up to 12 months
Muscle strength, measured by respiratory mouth pressure measurement, maximum inspiratoire mouthpressure, (Pimax) | up to 12 months
arterial inflammation as revealed by 18F-FDG PET . Standardized quantification parameters will be applied: Standardized uptake value (SUV), target-to-background ratio (TBR), most diseased segment analysis | up to 12 months
Calcification score of the coronary artery and thoracic aorta. The calcification will be quantified by using fully automated scoring and graded according to the Agatston score method | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, PhD., Principal Investigator — MAASTRO-clinic (senior researcher); Bas Kietselaer, MD,Phd, Principal Investigator — AzM/MUMC (cardiologist); Judith van Loon, MD,PhD, Principal Investigator — MAASTRO-clinic (radiation oncologist); Philippe Lambin, Prof,MD,Phd, Principal Investigator — MAASTRO-clinic (radiation oncologist); Anne-Marie Dingemans, MD, PhD, Principal Investigator — MAASTRO-clinic (pulmonogist)
Locations (2):
- Netherlands (2):
  - MAASTRO clinic, Maastricht, Limburg
  - Maastricht University Medical Center, Maastricht, Limburg